CLINICAL TRIAL: NCT01269515
Title: Optional Immunomodulating Therapy and Improved Vaccination Responses by Adjuvant Administration of a Cyclooxygenase Type 2 Inhibitor in Antiretroviral naïve HIV-infected Patients and Patients on ART
Brief Title: Immunomodulating Therapy and Improved Vaccination Responses by Cox-2 Inhibitor in HIV-infected Patients
Acronym: OUSCOX2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dag Kvale (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor-Investigator, Dag Kvale, Professor, Senior consultant, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OUSCOX2
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: HIV
Keywords: Cox-2 inhibitor; HIV; immune activation; immune modulating; progression markers; vaccine
MeSH Terms: interventions — Etoricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Etoricoxib 90 mg qd for 25 weeks ART- (Active Comparator): Etoricoxib for 25 weeks. Vaccination (Tetanus Toxoid, conjugated pneumococcal, seasonal influenza) after 5 weeks.
  Interventions: Drug: Etoricoxib
- Etoricoxib 90 mg qd for 2 weeks ART- (Active Comparator): Etoricoxib for 2 weeks. Vaccination (Tetanus Toxoid, conjugated pneumococcal, seasonal influenza) after 1 week.
  Interventions: Drug: Etoricoxib
- Control ART- (No Intervention): No Etoricoxib. Vaccination (Tetanus Toxoid, conjugated pneumococcal, seasonal influenza) after 1 week.
- Etoricoxib 90 mg qd for 25 weeks ART+ (Active Comparator): Etoricoxib for 25 weeks. Vaccination (Tetanus Toxoid, conjugated pneumococcal, seasonal influenza) after 5 weeks.
  Interventions: Drug: Etoricoxib
- Etoricoxib 90 mg qd for 2 weeks ART+ (Active Comparator): Etoricoxib for 2 weeks. Vaccination (Tetanus Toxoid, conjugated pneumococcal, seasonal influenza) after 1 week.
  Interventions: Drug: Etoricoxib
- Control ART+ (No Intervention): No Etoricoxib. Vaccination (Tetanus Toxoid, conjugated pneumococcal, seasonal influenza) after 1 week.

INTERVENTIONS:
Drug: Etoricoxib — 90 mg QD
  Other Names: Arcoxia
  Arms: Etoricoxib 90 mg qd for 2 weeks ART+; Etoricoxib 90 mg qd for 2 weeks ART-; Etoricoxib 90 mg qd for 25 weeks ART+; Etoricoxib 90 mg qd for 25 weeks ART-

SUMMARY:
Chronic immune activation is a central feature of HIV-infection, and the degree of activated T-cells is a better predictor of disease progression and mortality than plasma viral load. The study hypothesis is that the anti-inflammatory substance etoricoxib will dampen chronic immune activation and improve the effect of T-cell dependent vaccines in HIV-1 infected patients.

The aim of the present study is to explore the efficacy of the study drug on markers of immune activation and vaccine responses, as well as safety of the study drug, in HIV-infected patients not receiving antiretroviral therapy and in patients on long-term effective ART who had CD4 counts < 500.

DETAILED DESCRIPTION:
The current trial was based on our observations that augmented levels of cyclic adenosine monophosphate (cAMP) contribute to the T cell dysfunction in HIV-infected patients. In T cells, cAMP triggers a protein kinase A (PKA) - Csk - Lck inhibitory pathway that inhibits the proximal T cell receptor (TCR) signaling events. This mechanism may also be involved in the inhibitory function of regulatory T cells.

The investigators have hypothesized that elevated levels of cAMP in T cells from HIV-infected individuals result from increased production of prostaglandin E2 (PGE2) following activation-induced expression of cyclooxygenase type 2 (COX-2) in lymphoid tissues. Although the investigators have identified even COX-2 positive T cells in HIV-infected individuals, activated monocytes may be the major source of PGE2; high levels of COX-2 are produced de novo after a number of stimuli, particularly lipopolysaccharide (LPS). Circulating LPS is indeed increased in untreated chronic HIV infection due to enhanced translocation of microbial material and correlates to chronic immune activation and disease progression.

In three preceding clinical explorative trials, the investigators have demonstrated that COX-2 inhibition by COX-2 inhibitors (COX-2i) improves the immune functions of HIV patients, the first two studies included patients on antiretroviral treatment (ART). In the third trial the investigators also showed for the first time that treatment with a COX-2i was able to downregulate chronic immune activation and improve T cell functions (efficacy of T cell-dependent vaccine) in asymptomatic HIV-infected patients who did not use ART. In these patients, chronic immune activation was dampened as demonstrated; CD38 density on CD8+ T cells (primary endpoint) decreased by 24% by study week 12. This reduction could be extrapolated to a possible improvement of CD4+ T cell loss with 30 CD4 cells per ul per year with an approximate mean CD4 loss of 60 per ul per year. These data founded the basis for further support to this study through the GLOBVAC call program under the Norwegian Research Council (granted application for the current study).

ELIGIBILITY:
Inclusion Criteria:

ART- group: Confirmed diagnosis of HIV infection < 8 years prestudy

* no HIV-related clinical manifestations including acute HIV infection
* no current indication or use for antiretroviral treatment
* CD4+ count > 350 x 10^6 /l
* HIV RNA > 2000 copies/ml

ART+ group: Confirmed diagnosis of HIV infection

* no HIV-related clinical manifestations including acute HIV infection
* On stabile effective antiretroviral treatment (HIV RNA <50 copies/ml)
* CD4+ count < 500 x 10^6 /l
* HIV RNA > 2000 copies/ml

Exclusion Criteria:

* concomitant or sporadic use of NSAID, corticosteroids or other immune modulating therapies including interferon-alpha
* cholesterol > 7 M
* under treatment for hypertension or antihypertensive treatment indicated at inclusion
* cardiovascular events or stroke in parents, siblings or off-springs occurring < 55 years of age
* elevated serum creatinine
* diabetes type I or II
* known hypersensitivity for etoricoxib, capsule substances or sulphonamides
* active peptic ulcer or gastrointestinal haemorrhage
* history of asthma, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria or other allergic reactions after taking acetyl salicylic acid or NSAID including COX-2 inhibitors
* pregnancy or insufficient birth control for females
* breastfeeding
* seriously deranged liver function
* creatine clearance < 30 ml/min
* inflammatory bowel disease
* heart failure (NYHA II-IV)
* established ischaemic heart disease, peripheral arteriosclerosis and/or cerebrovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes in progression markers and vaccine responses within and between ART groups | After 6 months
  Changes in CD38 density (CD38 molecules per CD38+CD8+CD3+ T cells) and in humoral and cellular immune responses to study-specific vaccines.
Serious adverse events | During the 6 months study period
  Reductions of etoricoxib dose or stop of drug, adverse events including cardiovascular events, blood pressure, clinical chemistry.

SECONDARY OUTCOMES:
Changes in HIV Gag CD8+ T cell responses within and between ART groups | 6 months
  Changes in HIV Gag CD8+ T cell responses within and between ART groups
Changes in plasma markers of inflammation, coagulation and tryptophan metabolism within and between ART groups | 6 months
  Changes in plasma markers of inflammation, coagulation and tryptophan metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Dag Kvale, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Department of Infectious Diseases, Oslo University Hospital, Oslo
  - The Biotechnology Centre, University of Oslo, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Prebensen C, Troseid M, Ueland T, Dahm A, Sandset PM, Aaberge I, Waalen K, Dyrhol-Riise AM, Tasken K, Kvale D. Immune activation and HIV-specific T cell responses are modulated by a cyclooxygenase-2 inhibitor in untreated HIV-infected individuals: An exploratory clinical trial. PLoS One. 2017 May 2;12(5):e0176527. doi: 10.1371/journal.pone.0176527. eCollection 2017. PMID 28464042